CLINICAL TRIAL: NCT02756559
Title: MiRNAs Evaluating Lymphocyte Proliferation and Apoptosis as Well as Prognosis of Sepsis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Lixin Xie (Other)
Responsible Party: Sponsor-Investigator, Lixin Xie, Clinical Professor, Chinese PLA General Hospital
Organization: Chinese PLA General Hospital (Other)
Other Study IDs: S2015-068-01
Record Dates: First submitted 2016-04-25; First posted 2016-04-29 (Estimated); Last update posted 2016-05-02 (Estimated); Status verified 2016-04

CONDITIONS: T Lymphocyte Disorder
Keywords: sepsis; microRNAs
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- sepsis, severe sepsis and septic shock: Septic patients were divided into sepsis, severe sepsis and septic shock

SUMMARY:
Sepsis is a systemic inflammatory reaction caused by infection, trauma, etc. In the process of sepsis, the apoptosis of lymphocyte serves as a vital factor of immune dysfunction. Micro-RNAs (miRNAs) are endogenous small non-coding RNA molecules. Our previous studies have showed the diagnostic and prognostic value of a series circulant miRNAs in human serum in sepsis. The present research further study the regulatory mechanism of those miRNAs in lymphocyte in sepsis. Our research is based on the clinical value of miR-223, miR-15a, miR-16. The investigators discuss the potential role of miR-223, miR-15a, miR-16 in regulating the proliferation and apoptosis of lymphocyte in sepsis and aim to find new targets for sepsis treatment.

DETAILED DESCRIPTION:
Blood samples were collected from the Chinese People's Liberation Army General Hospital. The investigators collected samples in emergency intensive care unit (EICU), surgical intensive care unit (SICU) and respiratory intensive care unit (RICU) between July 2014 to March 2015. Septic patients were divided into sepsis, severe sepsis and septic shock according to the diagnostic criteria. Peripheral white blood cells were sorted into monocytes, lymphocytes and neutrophils by using flow cytometry (Flow Cytometry, FCM). Jurkat T cell lines were purchased from Chinese Academy of Medical Sciences Institute of basic medical sciences. miRNAs agomirs and antagonists were used to establish miR-223, miR-15a, miR-16 overexpression and knock-out transient transfection cell lines. Western blot was used to detect difference expression of protein expression.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Sepsis
* Agree with this study

Exclusion Criteria:

* Age <18 years
* Died within 24 hours
* Combined with HIV infection
* Agranulocytosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Blood samples were collected from the Chinese People's Liberation Army General Hospital. The investigators collected samples in emergency intensive care unit (EICU), surgical intensive care unit (SICU) and respiratory intensive care unit (RICU),within 24 hours admitted into ICU.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2014-01; Primary Completion 2017-06 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
all cause mortality | 28 days after admitted to ICU

CONTACTS AND LOCATIONS:
Overall Officials: Lixin Xie, Clinical Professor, Study Chair — Chinese PLA General Hospital
Locations (1):
- Chinese People's Liberation Army General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided